CLINICAL TRIAL: NCT00373503
Title: Effect of Lofexidine and Oral THC on Marijuana Withdrawal and Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 4942; R01DA019239 (NIH)
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Marijuana Dependence
Keywords: Lofexidine; Oral THC; Cannabinoids
MeSH Terms: conditions — Marijuana Abuse | interventions — lofexidine; Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- lofexidine, dronabinol, marijuana (Experimental): lofexidine (.6 mg qid), dronabinol (20 mg tid)
  Interventions: Drug: Lofexidine; Drug: dronabinol; Drug: Marijuana

INTERVENTIONS:
Drug: Lofexidine — alpha 2 adrenergic agonist, hypothesized to decrease noradrenergic activity
  Other Names: Britlofex
Drug: dronabinol — cannabinoid agonist hypothesized to decrease MJ withdrawal
  Other Names: THC
Drug: Marijuana — marijuana intoxication, withdrawal and relapse assessed
  Other Names: cannabis

SUMMARY:
The purpose of this study is to investigate the interaction between marijuana and two potential treatment medications: lofexidine and oral THC, with the direct goal of using this information to improve marijuana treatment outcome.

DETAILED DESCRIPTION:
Only a small percentage of dependent-marijuana smokers who are seeking treatment for their marijuana use is able to achieve sustained abstinence. The objective of this study is to investigate the interaction between marijuana and two potential treatment medications: lofexidine and oral THC, with the direct goal of using this information to improve marijuana treatment outcome. In mice, the α2-receptor agonist, clonidine, reversed symptoms of cannabinoid withdrawal (Lichtman et al., 2001). The purpose of this study is to determine if lofexidine, an α2-receptor agonist with a more favorable side-effect profile than clonidine, decreases symptoms of marijuana withdrawal and thus decreases marijuana relapse, as compared to placebo. Oral THC is FDA-approved for appetite enhancement. Lofexidine, which is currently not FDA-approved, is used in Europe to treat symptoms of heroin withdrawal, and to treat hypertension. For the purposes of this model, relapse is defined to a return to marijuana use after a period of abstinence. We have shown that oral THC reduces symptoms of marijuana withdrawal at doses that produce minimal intoxication (Haney et al., 2004). Thus, the effects of oral THC alone and in combination with lofexidine will be determined. The study will utilize an inpatient/outpatient, counter-balanced design, with each participant maintained on each of four medication conditions for 8 days each: placebo, lofexidine, oral THC, and oral THC combined with lofexidine. During the inpatient study phases, participants will have the opportunity to self-administer placebo or active marijuana 6 times per day. Outpatient phases are for medication clearance so no medications will be administered. This study will provide important information of the effect of these potential treatment medications on both marijuana withdrawal symptoms, and on subsequent marijuana self-administration.

ELIGIBILITY:
Inclusion Criteria:

* Current marijuana use: average of 3 marijuana cigarettes at least 4 times per week for the past 4 weeks
* Able to perform study procedures
* 21-45 years of age
* Women practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD)

Exclusion Criteria:

* Current, repeated illicit drug use (other than marijuana)
* Presence of significant medical illness (e.g., diabetes, cardiovascular disease, hypertension, clinically significant laboratory abnormalities)
* Bradycardia (55 beats/minute), hypotension (< 90 mmHg) including orthostatic hypotension (> 20 mmHg decrease in SP, or > 10 mmHg decrease in DP upon standing
* History of heart disease
* Request for drug treatment
* Current parole or probation
* Pregnancy or current lactation
* Recent history of significant violent behavior
* Major current Axis I psychopathology (e.g., major depressive disorder, bipolar disorder,suicide risk, schizophrenia)
* Current use of any prescription or over-the-counter medication

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
marijuana relapse | 4 days

SECONDARY OUTCOMES:
marijuana withdrawal symptoms | 3 days

OTHER OUTCOMES:
cardiovascular effects | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States